CLINICAL TRIAL: NCT01356901
Title: Persistence, Adherence and Clinical Effectiveness in Patients With Chronic Hepatitis B Viral Infection Treated With Entecavir in Real Life
Brief Title: Persistence, Adherence and Clinical Effectiveness of Entecavir in Chronic Hepatitis B Patients
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: AI463-232
Record Dates: First submitted 2011-04-15; First posted 2011-05-20 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-06

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment naïve and pre-treated CHB patients: subanalysis with migrant and non-migrant patients

SUMMARY:
The purpose of this observational study is to measure the real-life persistence, adherence and clinical effectiveness of entecavir in patients with chronic Hepatitis B viral infection.

DETAILED DESCRIPTION:
Sampling Method: Probability Sample (consecutive patient sampling)

ELIGIBILITY:
Inclusion Criteria:

* Male and female treatment naïve or pre-treated CHB patients of at least 18 years of age
* Written informed consent

Exclusion Criteria:

* All relevant conditions according to Summary of product characteristics (SmPC)
* Human immunodeficiency virus (HIV), Hepatitis C virus (HCV) or Hepatitis D virus (HDV) co-infection
* Patients currently included in any investigational trial on CHB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CHB Patients treated by Gastroenterologists/Hepatologists
Sampling Method: Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2011-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Chronic hepatitis B (CHB) patients treated with Entecavir (ETV) and any switch or add-on therapy who are persistent over a time period of two years in a real-life setting. | After 2 years
  A patient will be defined as non-persistent if he misses all his doses in more than 30 subsequent days or if he fails to show up at more than one subsequent visit.

SECONDARY OUTCOMES:
Adherence rates using administrative measures (continuous multiple-interval medication gaps, continuous single interval medication availability), and self-report measures, 8-item self-report Morisky Medication Adherence Scale (MMAS) | After 2 years
Reasons for therapy non-persistence (therapy discontinuation) and low therapy adherence (qualitative questionnaire for causal assessment of non-persistence/non-adherence) | After 2 years
Proportion of patients with HBV DNA below the limit of detection (according to local lab standard), mean log reduction of HBV DNA from baseline, proportion of subjects with normal ALT and with e antigen (eAg)/Surface antigen (sAg) seroconversion/loss | After 2 years
  Hepatitis B virus (HBV), desoxyribonucleic acid (DNA), Alanine aminotransferase (ALT)
Frequency of Serious adverse drug reaction ((S)ADR)s and study discontinuations due to (S)ADRs | After 2 years
Number of participants with occuring resistances based on results from resistance tests | After 2 years
Assessment of Health Status (SF-12® Health Survey) | Assessment of Health Status (SF-12 Health Survey) at year 1
Assessment of Health Status (SF-12® Health Survey) | Assessment of Health Status (SF-12 Health Survey) at year 2

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Herne, Germany

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx